CLINICAL TRIAL: NCT07249411
Title: In Vitro Oocyte Maturation With Autologous Exosomes in Women With Low Ovarian Reserve: Preliminary Phase of a Prospective Randomized Clinical Study
Brief Title: In Vitro Oocyte Maturation With Autologous Exosomes in Women
Acronym: Exosom2025-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotech Fertility C.A. (Other)
Responsible Party: Principal Investigator, Carmen Navarro, Reproductive Endocrinologist Consultant of Reproductive Medicine and Laparoscopic Surgery, Biotech Fertility C.A.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exosom2025-1
Record Dates: First submitted 2025-11-13; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Diminished Ovarian Reserve
Keywords: Oocyte maturation; Meiotic arrest; In vitro maturation; Autologous exosomes; Diminished ovarian reserve; Assisted reproductive technology

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled clinical trial designed to evaluate the safety and efficacy of the intervention in women diagnosed with infertility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI oocytes were cultured in conventional IVM medium supplemented with 10 µg of autologous exosomes o (Active Comparator): * Group I (Control): MI oocytes were cultured exclusively in conventional IVM medium (VITROLIFE®).
  * Group II (Experimental): MI oocytes were cultured in conventional IVM medium supplemented with 10 µg of autologous exosomes obtained using the ExoSMarT® exosome filtration system
  Interventions: Other: MI oocytes were cultured in conventional IVM medium supplemented with 10 µg of autologous exosomes obtained using the ExoSMarT® exosome filtration system
- MI oocytes were cultured exclusively in conventional IVM medium (VITROLIFE®). (Active Comparator): MI oocytes were cultured exclusively in conventional IVM medium (VITROLIFE®).
  Interventions: Other: MI oocytes were cultured in conventional IVM medium supplemented with 10 µg of autologous exosomes obtained using the ExoSMarT® exosome filtration system

INTERVENTIONS:
Other: MI oocytes were cultured in conventional IVM medium supplemented with 10 µg of autologous exosomes obtained using the ExoSMarT® exosome filtration system — MI oocytes were cultured in conventional IVM medium supplemented with 10 µg of autologous exosomes obtained using the ExoSMarT® exosome filtration system

SUMMARY:
This study is a preliminary, prospective, randomized, controlled clinical trial designed to evaluate the safety and feasibility of supplementing in vitro maturation (IVM) media with autologous exosomes in women with diminished ovarian reserve undergoing assisted reproductive technology. The purpose of the study is to determine whether autologous exosomes can support the meiotic progression of immature metaphase I oocytes during a 24-36 hour culture period and to establish whether the intervention is safe, biologically feasible, and suitable for further clinical evaluation. Mature oocytes obtained after culture are fertilized using intracytoplasmic sperm injection, and resulting embryos are cryopreserved for future transfer in a subsequent phase of the research. No embryo transfer is performed during this preliminary phase.

DETAILED DESCRIPTION:
Women with diminished ovarian reserve frequently present a high proportion of immature oocytes after controlled ovarian stimulation. These immature oocytes cannot be fertilized and limit the number of mature oocytes available for assisted reproductive procedures. Oocyte maturation is regulated by a coordinated set of intracellular signaling pathways, intercellular communication with granulosa cells, and molecular mechanisms that maintain meiotic arrest and trigger meiotic resumption. Emerging scientific evidence indicates that extracellular vesicles, including autologous exosomes, may play a role in supporting oocyte maturation through the transfer of bioactive molecules.

This preliminary clinical study was designed to evaluate the safety and feasibility of using autologous exosomes as a supplement to conventional in vitro maturation (IVM) media. The study population includes women aged 38-46 years with documented diminished ovarian reserve who declined oocyte donation and who met predefined clinical, endocrine, and reproductive criteria. All participants provided written informed consent. The study was conducted in accordance with national regulations and international ethical principles for research involving human subjects.

Eligible participants undergo controlled ovarian stimulation using recombinant follicle-stimulating hormone, human menopausal gonadotropin, and an antagonist protocol, followed by human chorionic gonadotropin triggering and oocyte retrieval. Only metaphase I oocytes are included in the intervention portion of the study. After identification, metaphase I oocytes are randomly assigned to one of two groups using a simple computer-generated randomization method.

In the control group, oocytes are cultured in conventional in vitro maturation medium. In the experimental group, oocytes are cultured in the same medium supplemented with a standardized quantity of autologous exosomes isolated from each participant according to the study protocol. Culture duration ranges from 24 to 36 hours. After the culture period, oocytes reaching metaphase II are fertilized via intracytoplasmic sperm injection to standardize the fertilization procedure. Embryos developing after fertilization are cultured under standardized laboratory conditions, evaluated according to established morphological criteria, and cryopreserved for use in a future phase of the research. Embryo transfer is not performed during this preliminary phase.

The primary objective of the study is to assess whether autologous exosome supplementation is feasible and safe for use in IVM culture systems. Secondary objectives include documenting the procedures involved in oocyte handling, fertilization, and embryo cryopreservation to support future phases of the study. The study does not include analysis of results or clinical outcomes, as no outcomes are permitted to be reported in the Protocol Section of the ClinicalTrials.gov record. A subsequent phase of the research will evaluate implantation, clinical pregnancy, and live birth after transfer of cryopreserved embryos generated in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Women with primary or secondary infertility associated with diminished ovarian reserve, defined by ultrasound findings and laboratory parameters (FSH > 10 mIU/mL and estradiol < 60 pg/mL).
* Serum anti-Müllerian hormone (AMH) concentration < 1 ng/mL.
* Antral follicle count < 3-6 follicles per ovary.
* Anatomical preservation of both ovaries.
* Body mass index (BMI) between 24.5 and 30 kg/m².
* Absence of active oncological pathologies or connective tissue diseases (collagenopathies).
* No history of clinically relevant hematological disorders.
* Adequate serum levels of vitamins essential for reproductive function, including vitamin D, B-complex, and vitamin C.
* Last live birth within ≤ 10 years prior to study initiation.
* Normal thyroid function (TSH and free thyroid hormones within range).
* Absence of antiphospholipid antibody syndrome.
* Male partner with semen parameters within normal limits, according to the World Health Organization (WHO) criteria, 2010 (5th edition) and 2021 (6th edition).
* Signed informed consent for participation in the study.

Exclusion Criteria:

* • Patients without a diagnosis of infertility.

  * Women without documented diminished ovarian reserve.
  * Serum anti-Müllerian hormone (AMH) concentration > 1 ng/mL.
  * Antral follicle count > 3-6 follicles per ovary.
  * Absence of one or both ovaries.
  * Body mass index (BMI) > 30 kg/m².
  * Presence of active oncological pathologies or connective tissue diseases (collagenopathies).
  * History of clinically relevant hematological disorders.
  * Deficient or altered serum levels of vitamins essential for reproductive function (vitamin D, B-complex, and vitamin C).
  * Last live birth > 10 years prior to study initiation.
  * Altered thyroid function (TSH or free thyroid hormones out of range).
  * History of antiphospholipid antibody syndrome.
  * Male partner with abnormal semen parameters according to the World Health Organization (WHO) criteria, 2010 (5th edition) and 2021 (6th edition).
  * Refusal to sign informed consent for study participation.

Ages: 38 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Proportion of Metaphase I Oocytes Reaching Metaphase II After In Vitro Cultureautologous exosomes obtained using the ExoSMarT® exosome filtration system | 24-36 hours
  This measure evaluates the number and proportion of metaphase I oocytes that progress to the metaphase II stage after 24-36 hours of in vitro culture in either conventional IVM medium or IVM medium supplemented with autologous exosomes. Maturation will be identified by the presence of the first polar body. Data will be summarized as a proportion of total metaphase I oocytes cultured.
Number of Mature Oocytes Fertilized After Intracytoplasmic Sperm Injection (ICSI) | Approximately 18 hours after ICSI
  This measure records the number and proportion of in vitro-matured metaphase II oocytes that demonstrate normal fertilization after ICSI, defined by the presence of two pronuclei under standard embryology laboratory criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotech Fertility C.A, Caracas, Venezuela

IPD SHARING:
Plan to Share IPD: No
Not but the individual participant data (IPD) from this study will be available to other qualified researchers upon reasonable request. Data sharing will be granted after a formal email request specifying the investigator's identity, institutional affiliation, and research objective. Access will be provided only for scientifically justified purposes, in compliance with confidentiality agreements and ethical standards protecting participant privacy.

REFERENCES:
- [Background] Mehlmann LM. Stops and starts in mammalian oocytes: recent advances in understanding the regulation of meiotic arrest and oocyte maturation. Reproduction. 2005 Dec;130(6):791-9. doi: 10.1530/rep.1.00793. PMID 16322539
- [Background] Chand AL, Legge M. Amino acid transport system L activity in developing mouse ovarian follicles. Hum Reprod. 2011 Nov;26(11):3102-8. doi: 10.1093/humrep/der298. Epub 2011 Sep 13. PMID 21914669
- [Background] Dupont S, Krust A, Gansmuller A, Dierich A, Chambon P, Mark M. Effect of single and compound knockouts of estrogen receptors alpha (ERalpha) and beta (ERbeta) on mouse reproductive phenotypes. Development. 2000 Oct;127(19):4277-91. doi: 10.1242/dev.127.19.4277. PMID 10976058
- [Background] Kiyama R, Wada-Kiyama Y. Estrogenic endocrine disruptors: Molecular mechanisms of action. Environ Int. 2015 Oct;83:11-40. doi: 10.1016/j.envint.2015.05.012. Epub 2015 Jun 11. PMID 26073844
- [Background] Coticchio G, Dal Canto M, Mignini Renzini M, Guglielmo MC, Brambillasca F, Turchi D, Novara PV, Fadini R. Oocyte maturation: gamete-somatic cells interactions, meiotic resumption, cytoskeletal dynamics and cytoplasmic reorganization. Hum Reprod Update. 2015 Jul-Aug;21(4):427-54. doi: 10.1093/humupd/dmv011. Epub 2015 Mar 4. PMID 25744083
- [Background] Esbert M, Reig A, Ballestros A, Seli E. Oocyte maturation defect in women undergoing IVF: contributing factors and effects on mature sibling oocyte outcomes. J Assist Reprod Genet. 2025 Mar;42(3):773-780. doi: 10.1007/s10815-024-03353-w. Epub 2025 Jan 9. PMID 39786528
- [Background] Coticchio G, Cimadomo D, Rienzi L. The daunting goal to rescue oocytes collected immature in conventional ovarian stimulation cycles. Fertil Steril. 2025 May;123(5):747-748. doi: 10.1016/j.fertnstert.2025.02.026. Epub 2025 Feb 22. PMID 39993495
- [Background] Navarro C, Torrecillas Cabrera P, Teppa Garran A. Comparative analysis of the use of autologous exosomes and platelet-derived growth factors in women with premature ovarian insufficiency and infertility: A prospective, randomized, observational, analytical study. Regen Ther. 2025 Jun 30;30:309-320. doi: 10.1016/j.reth.2025.06.007. eCollection 2025 Dec. PMID 40678344
- [Background] Tornell J, Billig H, Hillensjo T. Resumption of rat oocyte meiosis is paralleled by a decrease in guanosine 3',5'-cyclic monophosphate (cGMP) and is inhibited by microinjection of cGMP. Acta Physiol Scand. 1990 Jul;139(3):511-7. doi: 10.1111/j.1748-1716.1990.tb08953.x. PMID 2173353
- [Background] Cho WK, Stern S, Biggers JD. Inhibitory effect of dibutyryl cAMP on mouse oocyte maturation in vitro. J Exp Zool. 1974 Mar;187(3):383-6. doi: 10.1002/jez.1401870307. No abstract available. PMID 4362350
- [Background] Dekel N, Beers WH. Development of the rat oocyte in vitro: inhibition and induction of maturation in the presence or absence of the cumulus oophorus. Dev Biol. 1980 Mar 15;75(2):247-54. doi: 10.1016/0012-1606(80)90160-8. No abstract available. PMID 6154623
- [Background] Schultz RM, Montgomery RR, Belanoff JR. Regulation of mouse oocyte meiotic maturation: implication of a decrease in oocyte cAMP and protein dephosphorylation in commitment to resume meiosis. Dev Biol. 1983 Jun;97(2):264-73. doi: 10.1016/0012-1606(83)90085-4. PMID 6189752
- [Background] Horner K, Livera G, Hinckley M, Trinh K, Storm D, Conti M. Rodent oocytes express an active adenylyl cyclase required for meiotic arrest. Dev Biol. 2003 Jun 15;258(2):385-96. doi: 10.1016/s0012-1606(03)00134-9. PMID 12798295
- [Background] Hinckley M, Vaccari S, Horner K, Chen R, Conti M. The G-protein-coupled receptors GPR3 and GPR12 are involved in cAMP signaling and maintenance of meiotic arrest in rodent oocytes. Dev Biol. 2005 Nov 15;287(2):249-61. doi: 10.1016/j.ydbio.2005.08.019. Epub 2005 Oct 17. PMID 16229830
- [Background] Kovanci E, Rohozinski J, Simpson JL, Heard MJ, Bishop CE, Carson SA. Growth differentiating factor-9 mutations may be associated with premature ovarian failure. Fertil Steril. 2007 Jan;87(1):143-6. doi: 10.1016/j.fertnstert.2006.05.079. Epub 2006 Dec 6. PMID 17156781
- [Background] Vaccari S, Horner K, Mehlmann LM, Conti M. Generation of mouse oocytes defective in cAMP synthesis and degradation: endogenous cyclic AMP is essential for meiotic arrest. Dev Biol. 2008 Apr 1;316(1):124-34. doi: 10.1016/j.ydbio.2008.01.018. Epub 2008 Jan 26. PMID 18280465